CLINICAL TRIAL: NCT06123728
Title: The Clinical Application of Magnetocardiography (MCG) as a Non-invasive Diagnostic Tool for Evaluating Myocardial Ischemic Function in Patients With Stable Coronary Artery Disease
Brief Title: MCG is Clinically Applied to Evaluate Myocardial Ischemic Function in Patients With Stable Coronary Artery Disease
Status: Recruiting | Type: Observational
Sponsor: Nanhai Hospital, Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GJishen
Record Dates: First submitted 2023-10-21; First posted 2023-11-09 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Stable Coronary Artery Disease
Keywords: stable coronary artery disease; magnetocardiography; coronary CTA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this observational study is to evaluate the diagnostic effectiveness of magnetocardiography (MCG) in patients with stable coronary artery disease (SCAD) and compare it with coronary CTA (CCTA). Additionally, the study aims to determine the most suitable diagnostic index for MCG. The primary question it seeks to address is whether MCG or MCG combined with CCTA can be utilized to guide the clinical application of percutaneous coronary intervention (PCI) for coronary heart disease.

DETAILED DESCRIPTION:
1. Patients aged≥18 years with stable coronary artery disease (CCTA stenosis 30%-90%) underwent sequential examinations of MCG and CCTA. The results of CCTA were assessed using CT-FFR, and the diagnostic effectiveness of MCG in evaluating myocardial ischemia was analyzed using CT-FFR as the reference standard. Simultaneously, MCG was compared to CCTA to determine the clinical value of MCG in the functional evaluation of myocardial ischemia.
2. Coronary angiography was performed in patients who met the criteria for the procedure, and revascularization was carried out based on the intraoperative situation. Patients who underwent revascularization were followed up for 1 year, with major adverse cardiovascular events (MACE) as the endpoint. The clinical value of MCG in guiding the treatment of patients with SCAD was evaluated by reviewing the proportion of coronary angiography, revascularization, and MACE in the enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. Stable coronary artery disease patients with a coronary CTA stenosis degree of 30% to 90%.
3. Sign informed consent.

Exclusion Criteria:

1. Patients diagnosed with acute coronary syndrome.
2. Patients diagnosed with hypertrophic cardiomyopathy.
3. Patients diagnosed with dilated cardiomyopathy.
4. Patients with complex arrhythmias, such as frequent atrial premature beats, ventricular premature beats, and complete bundle branch block.
5. Patients with a left ventricular ejection fraction less than 50%.
6. Patients with chronic obstructive pulmonary disease, heart failure, kidney failure, or other serious diseases.
7. Pregnant women.
8. Patients with an allergy to contrast agents.
9. The study subjects who have metal grafts that interfere with magnetic cardiogram examination.
10. The study subjects who are unable to cooperate with magnetocardiogram examination and CTA.
11. Patients who have undergone coronary artery bypass grafting.
12. There are significant artifacts present in coronary CTA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected stable coronary artery disease were enrolled in a consecutive group at Nanhai Hospital of Guangdong Provincial People's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Consistency in comparing MCG and CT-FFR | 1 year
  Initially, MCG was conducted on each patient to assess the extent of myocardial ischemia using magnetic field distribution, pseudo-current density distribution, magnetic field intensity time spectrum line, and magnetic couple parameters. Simultaneously, the CT-FFR cut-off value of 0.8 was employed as the benchmark for this study. The agreement, sensitivity, specificity, and positive/negative predictive value of cardiac ischemia were compared between MCG and CT-FFR.

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 1 year
  Firstly, we performed coronary angiography in the above patients who met the indications of coronary angiography and performed revascularization according to the intraoperative conditions. The revascularized patients were then followed up for 1 year with major adverse cardiovascular events as the endpoint. By reviewing the ratio of coronary angiography, revascularization, and incidence of MACE in enrolled patients, the value of MCG in guiding the clinical treatment of patients with stable coronary disease was evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanhai Hospital, Guangdong Provincial People's Hospital, Foshan, Guangdong, China